CLINICAL TRIAL: NCT07189091
Title: Effect of Reduced Sodium Chloride in Fluid Creep and Maintenance Fluids in Critically Ill Adults: A Randomized Controlled Trial
Brief Title: CReep and Maintenance flUid Sodium Chloride ADministration rEduction in cRitically Ill adultS
Acronym: CRUSADERS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Ziekenhuis aan de Stroom (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Edge 003813; 2025-520744-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: Critical Care, Intensive Care; Fluid Accumulation; Fluid and Electrolyte Imbalance; Critical Illness; Fluid Balance Outcomes
Keywords: Intensive Care Unit; Critically Ill; Critical Illness; Intravenous fluids; Maintenance fluids; Fluid Creep; Sodium chloride reduction; Salt reduction; Hypotonic fluids; Saline (NaCl 0.9%); Fluid balance; Electrolyte disorders; Glycemic control; Acute kidney injury; Mechanical ventilation; Organ support; Hyponatremia
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Hyponatremia | interventions — Glucose; Saline Solution; Plasmalyte A

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, multicenter, randomized, double-blind, parallel-group phase IV trial conducted in four mixed ICUs in Belgium. Adult patients expected to require prolonged ICU care are randomized 1:1 to a sodium-chloride reduction strategy (NaCl-poor arm) or to a standard isotonic fluid strategy (NaCl-rich arm). Randomization is stratified by study site, surgical admission, and invasive mechanical ventilation at enrollment, using permuted blocks with concealed allocation. Each study arm consists of two components: composition of fluid creep (diluents and line patency solutions) and composition of maintenance fluids. All fluids are market-authorized products prepared and blinded by hospital pharmacy, supplied in opaque bags labeled only with trial codes. The assigned strategy is maintained throughout the ICU stay or until blinded study fluids are no longer available under the rotating allocation schedule. Follow-up continues until day 90 after ICU admission
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is ensured by the use of opaque blinding labels applied by unblinded hospital pharmacists. These labels conceal the identity of the solution while leaving mandatory information such as fluid volume, batch number, and expiry date visible, in line with regulatory requirements. The fluids are otherwise indistinguishable and are labeled only with a randomization code letter. Randomization letters are changed monthly to prevent recognition of fluid composition. Only the pharmacists are unblinded; they handle labeling, storage, and distribution but are not involved in patient care or outcome assessment. In the ICU, nurses and physicians administer fluids documented simply as "study fluid," without access to the underlying composition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium chloride reduction strategy, the NaCl-poor arm (Active Comparator): Participants receive a sodium-chloride reduction strategy during their ICU stay. Medications are diluted in glucose 5% (unless another solvent is mandatory), and intravenous line patency fluids are glucose 5%. Daily maintenance fluids are NaCl 0.3% in glucose 3.3%, with the volume determined by the treating physician. The goal is to reduce sodium and chloride exposure while maintaining fluid and electrolyte support.
  Interventions:
  Drug: Glucose 5% Drug: NaCl 0.3% in Glucose 3.3%
  Interventions: Drug: Glucose 5% for fluid creep; Drug: NaCl 0.3% in glucose 3.3% as maintenance fluid
- Isotonic fluid strategy, the NaCl-rich arm (Active Comparator): Participants receive a standard isotonic fluid strategy during their ICU stay. Medications are diluted in NaCl 0.9% (unless another solvent is mandatory), and intravenous line patency fluids are NaCl 0.9%. Daily maintenance fluids are PlasmaLyte, with the volume determined by the treating physician. This reflects the common standard of care in many ICUs.
  Interventions:
  Drug: NaCl 0.9% Drug: PlasmaLyte
  Interventions: Drug: NaCl 0.9% (normal saline) for fluid creep; Drug: PlasmaLyte as maintenance fluid

INTERVENTIONS:
Drug: Glucose 5% for fluid creep — * Medications, including concentrated electrolytes, are dissolved in glucose 5% except when another solvent is mandatory according to the responsible pharmacist.
  * Infusions to keep intravenous lines open are glucose 5%
  Arms: Sodium chloride reduction strategy, the NaCl-poor arm
Drug: NaCl 0.9% (normal saline) for fluid creep — * Medications, including concentrated electrolytes, are dissolved in NaCl 0.9% except when another solvent is mandatory according to the responsible pharmacist.
  * All infusions to keep intravenous lines open are NaCl 0.9%.
  Arms: Isotonic fluid strategy, the NaCl-rich arm
Drug: PlasmaLyte as maintenance fluid — * Type: Maintenance fluid is PlasmaLyte. Potassium chloride or potassium phosphate can be added (or administered separately) whenever deemed necessary.
  * Rate: at the discretion of the treating physician, typically 25-30 ml/kg of body weight with a maximum of 100 ml/hour, accounting for concomitant fluid sources such as nutrition and fluid creep. It is allowed to prescribe a higher volume of study maintenance fluids to include replacement if both study fluids are considered appropriate.
  Arms: Isotonic fluid strategy, the NaCl-rich arm
Drug: NaCl 0.3% in glucose 3.3% as maintenance fluid — * Type: maintenance fluid is NaCl 0.3% in glucose 3.3%. Potassium chloride or potassium phosphate can be added (or administered separately) at the discretion of the treating physician whenever necessary.
  * Rate: at the discretion of the treating physician, typically 25-30 ml/kg of body weight with a maximum of 100 ml/hour, accounting for concomitant fluid sources such as nutrition and fluid creep. It is allowed to prescribe a higher volume of study maintenance fluids to include replacement if both study fluids are considered appropriate
  Arms: Sodium chloride reduction strategy, the NaCl-poor arm

SUMMARY:
This study is enrolling adult patients who require a prolonged stay in the intensive care unit (ICU). These patients often receive large amounts of intravenous fluids, which can contain more salt (sodium and chloride) than the body normally needs. Extra salt and water can build up in the body and may delay recovery.

The study will test two strategies:

Fluid creep: These are fluids used to dilute medications or keep intravenous lines open. Usually, the choice is based on habit. In the intervention group, a salt-free glucose 5% solution will be used (if the responsible pharmacist confirms it is compatible with the medication).

Maintenance fluids: These fluids cover daily needs for water and electrolytes. In the intervention group, a lower-salt solution (NaCl 0.3% in glucose 3.3%) will be given, with volume decided by the treating physician.

The comparison group will receive usual care: NaCl 0.9% (commonly called "normal saline") for fluid creep, and an isotonic solution (PlasmaLyte) for maintenance fluids.

The main outcome is the number of days patients are alive and free of life support (such as ventilator or dialysis) during the first 90 days. Other outcomes include abnormal sodium, chloride, or glucose levels, fluid balance and need for diuretics, kidney injury, use of dialysis, time on the ventilator, survival, and length of ICU and hospital stay.

A smaller substudy (SALADIN) will measure in detail how the body handles sodium, chloride, and water using additional calculation on blood tests, urine collections, body weight, and bioimpedance analysis

DETAILED DESCRIPTION:
Critically ill patients admitted to the intensive care unit (ICU) often receive large volumes of intravenous fluids. Beyond resuscitation fluids, which have been extensively studied, two other sources contribute substantially to fluid, sodium, and chloride exposure:

Fluid creep, the use of diluents and small-volume infusions to dissolve medications or maintain line patency.

Maintenance fluids, prescribed to cover daily fluid and electrolyte needs when oral intake is insufficient.

Together, fluid creep and maintenance fluids account for more than half of all intravenous fluids given in ICU patients. These fluids frequently contain supraphysiologic amounts of sodium and chloride. Because the kidneys of critically ill patients are unable to excrete these excesses efficiently, sodium and chloride accumulate, leading to positive fluid balances, electrolyte disturbances, pulmonary edema, renal dysfunction, and prolonged organ support. Observational data have linked both fluid overload and hyperchloremia to higher morbidity and mortality.

Prior research has focused mainly on resuscitation fluids. Large randomized trials comparing chloride-rich saline to balanced crystalloids demonstrated only small differences in outcomes, in part because resuscitation fluids make up a limited fraction of overall fluid exposure. In contrast, fluid creep and maintenance solutions offer a larger and modifiable source of sodium and chloride. Small studies and volunteer experiments have shown that sodium-poor maintenance fluids and sodium-free diluents reduce fluid retention and hyperchloremia, but their effect on patient-centered outcomes has never been tested in a large randomized trial.

CRUSADERS (CReep and maintenance flUid Sodium chloride ADministration Reduction in cRitically ill adultS) is a multicenter, randomized, double-blind, phase IV, low-intervention trial designed to address this evidence gap. The trial compares two strategies:

NaCl-poor arm (intervention):

Fluid creep: medications are dissolved in glucose 5% (except when another diluent is mandatory); line patency fluids are glucose 5%.

Maintenance fluids: NaCl 0.3% in glucose 3.3%, with volume determined by the treating physician.

NaCl-rich arm (control):

Fluid creep: medications are dissolved in NaCl 0.9%; line patency fluids are NaCl 0.9%.

Maintenance fluids: PlasmaLyte, with volume determined by the treating physician.

All study fluids are licensed, widely used hospital products. Blinding is achieved through repackaging into opaque study bags labeled only with trial codes. Treating teams decide indications and volumes, ensuring pragmatic applicability while isolating the effect of fluid composition.

The primary endpoint is days alive and without life support (DAWOLS) at 90 days after ICU admission, an outcome that integrates survival and duration of mechanical ventilation or renal replacement therapy. Secondary outcomes include electrolyte disorders (hyponatremia, hypernatremia, hyperchloremia), fluid balance and diuretic use, acute kidney injury, renal replacement therapy, mechanical ventilation, glycemic control, mortality, and ICU/hospital length of stay. Exploratory outcomes include biochemical markers of salt-induced catabolism such as the serum urea-to-creatinine ratio.

A nested substudy (SALADIN - SAlt baLAnce Detailed INsight) will provide mechanistic insights into sodium, chloride, and water handling. In this subgroup, detailed daily balances will be calculated from fluid intake and 24-hour urine collections, combined with measurements of free water clearance, bioelectrical impedance analysis, body weight, and volume kinetics modeling.

The trial will recruit 640 adult ICU patients across four Belgian mixed ICUs. Inclusion requires expected ICU stay >48 hours and anticipated exposure to maintenance fluids or significant fluid creep. Patients with contraindications to hypotonic fluids, severe baseline hyponatremia, imminent death, chronic dialysis, or exclusive palliative/organ donation admission are excluded.

Patients are randomized 1:1 with stratification by site, mechanical ventilation, and surgical admission. Study treatment continues throughout the ICU stay or until study fluids are no longer available according to the blinded allocation schedule (minimum 28 days after randomization). Follow-up continues until 90 days after ICU admission.

The CRUSADERS trial is investigator-initiated, funded by the Research Foundation Flanders (FWO), and sponsored by Antwerp University Hospital. It is conducted under European Union (EU) Clinical Trial Regulation (536/2014) with central review via the Clinical Trial Information System (CTIS). Given the exclusive use of approved fluids in routine indications, the trial is classified as low-intervention. A Data and Safety Monitoring Board oversees safety with predefined stopping rules and interim analysis after half the planned population has been followed.

By targeting sodium and chloride in fluid creep and maintenance solutions rather than resuscitation fluids, CRUSADERS aims to test a simple, cost-neutral, and widely applicable strategy to improve survival and reduce life support dependence in critically ill patients. If positive, the trial may provide a strong evidence base for revising international fluid therapy guidelines and daily ICU practice.

ELIGIBILITY:
Inclusion criteria

1. At least 18 years of age
2. Patients who are admitted to the ICU for medical or surgical emergencies, including complications of elective surgery
3. The treating physician expects the patient will still require ICU care in two days, indicating a severe or complex condition at enrollment
4. The patient is expected to receive at least 300 mL of fluid creep or at least 1 liter of maintenance fluid according to study-arm during the first 24h after inclusion

Exclusion Criteria:

1. A contraindication to hypotonic fluids due to risk of brain edema (including traumatic brain injury, major stroke, intracranial/subarachnoid hemorrhage, meningoencephalitis, intracranial malignancies…), with the timing and clinical judgment left at the discretion of the treating physician.
2. Hyponatremia below 131 mmol/L at admission
3. Admission solely for treatment of fluid accumulation due to cardiac decompensation, without other acute medical conditions requiring ICU-level care. Note: Patients with heart failure as a comorbidity, those on chronic diuretic therapy, or presenting with edema/bilateral lung infiltrates due to other conditions (e.g., sepsis, pneumonia) are not excluded.
4. Patient's death is deemed imminent and inevitable, admission for palliative care or admission solely for organ donation
5. Patient receiving chronic renal replacement therapy
6. Patients referred after a stay of more than 24 hours in another ICU
7. Patients randomized in CRUSADERS before
8. Patient is co-enrolled in an unapproved concomitant ICU-trial or in any trial with an intervention that affects fluid administration or fluid balance

Additional exclusion criteria for the SALADIN nested substudy

1. Patients expected to require renal replacement therapy within 24 hours
2. Increased insensible fluid losses: burns, extensive wounds or skin defects or massive diarrhea,…
3. Patients without a urine catheter
4. Patients expected to require bladder irrigation within 24 hours
5. Patients on chronic treatment with loop or thiazide diuretics (including combination preparations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Days alive and without life support at day 90 (DAWOLS90) | From admission until day 90 counted from ICU admission (= Day 1)
  The composite endpoint DAWOLS90 is defined as the number of days alive and without the use of life support within 90 days counted from ICU admission. Unit of measure: days. Patients who die before D90 are assigned zero days. The following life-support therapies are considered 1/ Mechanical ventilation: includes invasive and noninvasive ventilation, including continuous positive airway pressure (CPAP) but excluding high-flow nasal oxygen. Each ICU day counts as a ventilator day if support is in place. Post-extubation days are counted as ventilator-free only if no re-intubation occurs within 48 hours. 2/ Renal replacement therapy (RRT): includes continuous RRT, peritoneal dialysis, or intermittent hemodialysis (IHD). If IHD is given, periods with up to 3 days between sessions are counted as days with RRT.

SECONDARY OUTCOMES:
Occurrence of moderate and severe hyponatremia | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants with at least one episode of:
  Moderate hyponatremia: serum sodium 125-129 mmol/L Severe hyponatremia: serum sodium <125 mmol/L
  To be counted as an event, the sodium level must decrease by at least 3 mmol/L from baseline to reduce misclassification due to pre-existing mild hyponatremia or analytical variation. Assessments are based on daily routine morning serum sodium values from the central laboratory (ion-specific electrode). If available, paired serum albumin and point-of-care sodium values (measured within 2 hours) will be recorded to allow cross-checks and sensitivity analyses
Occurrence of moderate and severe hypernatremia | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants with at least one episode of:
  Moderate hypernatremia: serum sodium 151-155 mmol/L Severe hypernatremia: serum sodium >155 mmol/L
  To be counted as an event, the sodium level must increase by at least 3 mmol/L from baseline to account for pre-existing mild hypernatremia and analytical variation. Assessments are based on daily routine morning serum sodium values from the central laboratory (ion-specific electrode). If available, paired serum albumin and point-of-care sodium values (measured within 2 hours of the central measurement) will be recorded to allow cross-checks and sensitivity analyses.
Occurrence of moderate and severe hyperchloremia | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants with at least one episode of:
  Moderate hyperchloremia: serum chloride 111-115 mmol/L Severe hyperchloremia: serum chloride >115 mmol/L
  To be counted as an event, the chloride level must increase by at least 2 mmol/L from baseline to account for pre-existing mild hyperchloremia and analytical variation. Assessments are based on daily routine morning serum chloride values from the central laboratory (ion-specific electrode). If available, paired serum albumin and point-of-care chloride values (measured within 2 hours of the central measurement) will be recorded to allow cross-checks and sensitivity analyses
Time to first administration of intravenous loop diuretic | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the time (in hours) from randomization until the first administration of an intravenous loop diuretic (e.g., furosemide or bumetanide). The exact timestamp of first administration is recorded.
Proportion of ICU days with intravenous loop diuretic use | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of ICU days during which a participant receives at least one dose of an intravenous loop diuretic, expressed as a proportion of total ICU days.
Cumulative fluid balance in mL up to first IV loop diuretic use | From ICU admission until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the cumulative net fluid balance, excluding insensible losses. Daily fluid balance is calculated as total inputs minus total outputs (mL per ICU day).
  Inputs: study fluids, non-study fluid creep, non-study maintenance and replacement fluids, non-study resuscitation fluids, enteral and parenteral nutrition, blood products, and oral intake.
  Outputs: urine output, net ultrafiltration by renal replacement therapy, gastric aspirates, drain outputs, and diarrhea (if precisely measured).
  The cumulative fluid balance is the sum of all daily fluid balances from ICU admission until the morning of the first ICU day on which an intravenous loop diuretic is prescribed.
Occurrence of hyperglycemia | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the proportion of glucose measurements >180 mg/dL relative to the total number of glucose assessments during the ICU stay. Mean daily glucose values will also be calculated for each ICU day. Assessments are based on point-of-care blood gas analyzer values, which are routinely collected multiple times per day in all ICU patients.
Occurrence of hypoglycemia | From randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants with at least one episode of hypoglycemia, serum glucose <70 mg/dL, measured on routine point-of-care blood gas analysis. Severe hypoglycemia (<40 mg/dL) is separately recorded as a serious adverse reaction.
Occurrence of new-onset acute kidney injury (AKI) | From third ICU day after randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants who develop new-onset AKI stage 2 or 3 according to KDIGO criteria (Kidney Disease: Improving Global Outcomes), starting from the third ICU day after randomization. AKI classification is based on daily serum creatinine (central laboratory morning samples) and urine output collected every 12-24 hours. KDIGO stage 1 is not assessed in this trial.
Occurrence of new-onset need for renal replacement therapy (RRT) | From the second ICU day after randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants requiring new initiation of RRT (continuous renal replacement therapy, peritoneal dialysis, or intermittent hemodialysis). To attribute RRT to the intervention, only events starting on or after the second ICU day following randomization are considered.
Renal replacement therapy-free days at day 90 | From ICU admission until day 90 counted from ICU admission.
  Calculated as the number of days during the 90-day observation period that a participant is alive and not receiving renal replacement therapy (RRT). For intermittent hemodialysis, periods with up to 3 days between sessions are counted as days on RRT.
Occurrence of new-onset need for mechanical ventilation | From the second ICU day after randomization until ICU discharge (up to day 90 counted from ICU admission)
  Defined as the number of participants who newly require mechanical ventilation after randomization. Mechanical ventilation includes invasive and noninvasive ventilation (including continuous positive airway pressure (CPAP)) but excludes high-flow nasal oxygen. To attribute events to the intervention, only new initiation from the second ICU day after randomization is considered.
Ventilator-free days at day 90 | From ICU admission until ICU discharge (up to day 90 counted from ICU admission)
  Calculated as the number of days during the 90-day observation period that a participant is alive and free of mechanical ventilation. Mechanical ventilation includes invasive and noninvasive ventilation (including CPAP) but excludes high-flow nasal oxygen. Following extubation, days are counted as ventilator-free only if no re-intubation occurs within 48 hours.
Days alive and out of hospital at day 90 (DAOH90) | From ICU admission until day 90 counted from ICU admission.
  Defined as the number of days a participant is alive and outside the hospital during the 90 days after ICU admission. If a patient is discharged and later readmitted, both admissions are included in the total number of hospitalization days. Mortality is penalized and assigned a value of zero DAOH. DAOH is calculated at day 90 counted from ICU admission.
ICU length of stay | From ICU admission until ICU discharge (up to day 90 counted from ICU admission).
  Defined as the number of calendar days from ICU admission to ICU discharge, including referral or transfer to other ICUs following the same admission.
Hospital length of stay | From ICU admission until hospital discharge (up to day 90 counted from ICU admission)
  Defined as the number of calendar days from ICU admission to hospital discharge, including transfers to other hospitals. Discharges or transfers to rehabilitation wards within the same hospital are not counted as hospital length of stay.
ICU mortality | From ICU admission until discharge from the index ICU episode, including any continuous referrals/transfers to other ICUs (up to day 90 counted from ICU admission)
  Death occurring at any time while continuously in ICU during the index (initial) ICU episode. Inter-ICU transfers are considered part of the same continuous ICU episode. Deaths after discharge from the index ICU episode-whether on the ward or during any later ICU readmission within the same hospital admission-are not counted.
Hospital mortality | From ICU admission until discharge from the index hospital admission (up to day 90 counted from ICU admission)
  Death occurring at any time during the index (initial) hospital admission, irrespective of location (ICU or ward within the same hospital) and including transfers to other hospitals within the same continuous admission. Deaths after discharge from the index hospital admission are not counted, even if the patient is readmitted later.

OTHER OUTCOMES:
Daily sodium, chloride and glucose administration | From ICU admission until ICU discharge (up to day 90 counted from ICU admission).
  Total daily amount of sodium, chloride, and glucose (mmol or g per ICU day) from study fluids, non-study maintenance, replacement and resuscitation fluids, enteral and parenteral nutrition, and blood products (sodium/chloride content estimated from reference values). Excludes non-study fluid creep and oral intake.
Cumulative sodium, chloride and glucose administration | From ICU admission until ICU discharge (up to day 90 counted from ICU admission).
  Running total of sodium, chloride, and glucose (mmol or g) from ICU admission onward. Each day's administered amount is added to all previous ICU days. Same sources and exclusions as for daily administration.
Daily fluid balance (mL) | From ICU admission until ICU discharge, day 90 counted from ICU admission, removal of bladder catheter or initiation of bladder irrigation, whichever comes first.
  Daily fluid balance is calculated as inputs minus outputs (mL per ICU Day).
  Inputs: study fluids, non-study fluid creep, non-study maintenance and replacement fluids, non-study resuscitation fluids, enteral and parenteral nutrition, blood products, and oral intake.
  Outputs: urine output, net ultrafiltration by renal replacement therapy, gastric aspirates, drain outputs, and diarrhea (if precisely measured).
  From the time renal replacement therapy or intravenous loop diuretics are initiated, fluid balance will be analyzed separately from patients who do not receive these interventions.
Cumulative fluid balance (mL) | From ICU admission until ICU discharge, day 90 counted from ICU admission, removal of bladder catheter or initiation of bladder irrigation, whichever comes first.
  Cumulative fluid balance is defined as the running total of daily net fluid balances (inputs minus outputs), excluding insensible losses. Each day's balance is added to that of all previous ICU days, allowing assessment at any time during the ICU stay. Daily fluid balance is calculated as inputs minus outputs (mL per ICU Day).
  Inputs: study fluids, non-study fluid creep, non-study maintenance and replacement fluids, non-study resuscitation fluids, enteral and parenteral nutrition, blood products, and oral intake.
  Outputs: urine output, net ultrafiltration by renal replacement therapy, gastric aspirates, drain outputs, and diarrhea (if precisely measured).
  From the time renal replacement therapy or intravenous loop diuretics are initiated, fluid balance will be analyzed separately from patients who do not receive these interventions.
Serum urea-to-creatinine ratio | From the first morning after randomization until ICU discharge or initiation of RRT (up to day 90).
  Defined as the change in serum urea-to-creatinine ratio, measured every other ICU day starting the first morning after randomization in patients not receiving renal replacement therapy (RRT). Serum creatinine is assessed as part of routine care, and serum urea is measured from the same morning blood sample without additional sampling. Urea measurements are discontinued from the day RRT is initiated, and patients on RRT are excluded from this analysis. This endpoint is exploratory and based on the rationale that higher sodium exposure, as in the NaCl-rich arm, may increase muscle catabolism. The serum urea-to-creatinine ratio is an established biomarker of catabolism in critically ill patients.
Daily sodium and chloride balance (SALADIN substudy) | From ICU admission until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Net daily balance of sodium and chloride (mmol per ICU day), defined as inputs minus outputs.
  Inputs: study fluids, non-study maintenance and replacement fluids and resuscitation fluids, enteral and parenteral nutrition, and blood products (sodium/chloride content estimated from reference values). Excludes non-study fluid creep and oral intake.
  Outputs: sodium and chloride content of all urine collected during the ICU day Urine samples are performed until the ICU day on which bladder catheter removal, initiation of bladder irrigation, start of renal replacement therapy, or ICU discharge occurs, whichever comes first.
Cumulative sodium and chloride balance (SALADIN substudy) | From ICU admission until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Running total of daily sodium and chloride balances. Each day's balance is added to that of all previous ICU days, allowing assessment at any time during the ICU stay.
  Net daily balance of sodium and chloride (mmol per ICU day), defined as inputs minus outputs.
  Inputs: study fluids, non-study maintenance and replacement fluids and resuscitation fluids, enteral and parenteral nutrition, and blood products (sodium/chloride content estimated from reference values). Excludes non-study fluid creep and oral intake.
  Outputs: sodium and chloride content of all urine collected during the ICU day Urine samples are performed until the ICU day on which bladder catheter removal, initiation of bladder irrigation, start of renal replacement therapy, or ICU discharge occurs, whichever comes first.
Solute-free water clearance (SALADIN substudy) | From ICU admission until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Derived from urine and plasma osmolality and urine flow rate. Reported as mL per ICU day. Formula: Solute-free water clearance CH2O = V × (1 - Uosm/Posm), where V = urine flow rate, Uosm = urine osmolality, and Posm = plasma osmolality. Calculated daily during ICU stay in participants with 24-hour urine collections.
Electrolyte-free water clearance (SALADIN substudy) | From ICU admission until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Derived from urine sodium, urine potassium, plasma sodium, and urine flow rate. Reported as mL per ICU day. Formula Electrolyte-free water clearance: CeH2O = V × (1 - (UNa + UK)/PNa)), where V = urine flow rate, UNa = urine sodium concentration, UK = urine potassium concentration, and PNa = plasma sodium concentration.
  Calculated daily during ICU stay in participants with 24-hour urine collections.
Volume kinetics (SALADIN substudy) | From ICU admission until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Model-based analysis of administered fluid volumes and urine output to describe distribution and clearance of infused solutions. Performed in participants included in the SALADIN substudy with complete fluid and urine balance data.
Measured body weight (SALADIN substudy) | From ICU admission until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Daily body weight recorded in substudy participants to quantify changes in body fluid volume and tissue mass during critical illness.
Fluid distribution (BIA-derived) (SALADIN substudy) | From randomization until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Noninvasive bioelectrical impedance analysis (BIA) will be performed once daily up to every third ICU day in substudy participants using a multi-frequency analyzer. Fluid distribution parameters assessed include total body water, intracellular water, extracellular water, intravascular and extravascular distribution, and volume excess. Results are used to evaluate dynamic changes in fluid status during critical illness and to relate these to sodium and chloride balance.
Body Composition (BIA-derived) (SALADIN-substudy) | From randomization until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Noninvasive bioelectrical impedance analysis (BIA) will be performed once daily up to every third ICU day in substudy participants using a multi-frequency analyzer. Body composition parameters assessed include fat-free mass, fat mass, muscle mass, protein, mineral, and bone content. Serial measurements are used to assess changes in tissue composition over the course of critical illness.
Metabolic Indices (BIA-derived) (SALADIN substudy) | From randomization until ICU discharge or end of substudy sampling (up to day 90 counted from ICU admission)
  Noninvasive bioelectrical impedance analysis (BIA) will be performed once daily up to every third ICU day in substudy participants using a multi-frequency analyzer. Metabolic indices include resting metabolic rate, glycogen deposits, phase angle, and malnutrition index. These indices are evaluated to explore metabolic changes and nutritional status during critical illness, and their relationship with sodium and chloride balance.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Van Regenmortel, MD, PhD, Principal Investigator — Ziekenhuis aan de Stroom (ZAS) Network of Hospitals
Locations (4):
- Belgium (4):
  - ZAS Middelheim, Antwerp
  - ZAS Cadix, Antwerp
  - Antwerp University Hopsital (UZA), Edegem
  - ZAS Paflijn, Merksem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granholm A, Schjorring OL, Jensen AKG, Kaas-Hansen BS, Munch MW, Klitgaard TL, Crescioli E, Kjaer MN, Strom T, Lange T, Perner A, Rasmussen BS, Moller MH. Association between days alive without life support/out of hospital and health-related quality of life. Acta Anaesthesiol Scand. 2023 Jul;67(6):762-771. doi: 10.1111/aas.14231. Epub 2023 Mar 21. PMID 36915265
- [Background] Van Regenmortel N, Verbrugghe W, Roelant E, Van den Wyngaert T, Jorens PG. Maintenance fluid therapy and fluid creep impose more significant fluid, sodium, and chloride burdens than resuscitation fluids in critically ill patients: a retrospective study in a tertiary mixed ICU population. Intensive Care Med. 2018 Apr;44(4):409-417. doi: 10.1007/s00134-018-5147-3. Epub 2018 Mar 27. PMID 29589054
- [Background] Van Regenmortel N, Moers L, Langer T, Roelant E, De Weerdt T, Caironi P, Malbrain MLNG, Elbers P, Van den Wyngaert T, Jorens PG. Fluid-induced harm in the hospital: look beyond volume and start considering sodium. From physiology towards recommendations for daily practice in hospitalized adults. Ann Intensive Care. 2021 May 17;11(1):79. doi: 10.1186/s13613-021-00851-3. PMID 33999276
- [Background] Van Regenmortel N, Hendrickx S, Roelant E, Baar I, Dams K, Van Vlimmeren K, Embrecht B, Wittock A, Hendriks JM, Lauwers P, Van Schil PE, Van Craenenbroeck AH, Verbrugghe W, Malbrain MLNG, Van den Wyngaert T, Jorens PG. 154 compared to 54 mmol per liter of sodium in intravenous maintenance fluid therapy for adult patients undergoing major thoracic surgery (TOPMAST): a single-center randomized controlled double-blind trial. Intensive Care Med. 2019 Oct;45(10):1422-1432. doi: 10.1007/s00134-019-05772-1. Epub 2019 Oct 1. PMID 31576437
- [Background] Sakr Y, Vincent JL, Reinhart K, Groeneveld J, Michalopoulos A, Sprung CL, Artigas A, Ranieri VM; Sepsis Occurence in Acutely Ill Patients Investigators. High tidal volume and positive fluid balance are associated with worse outcome in acute lung injury. Chest. 2005 Nov;128(5):3098-108. doi: 10.1378/chest.128.5.3098. PMID 16304249
- [Background] Silversides JA, Major E, Ferguson AJ, Mann EE, McAuley DF, Marshall JC, Blackwood B, Fan E. Conservative fluid management or deresuscitation for patients with sepsis or acute respiratory distress syndrome following the resuscitation phase of critical illness: a systematic review and meta-analysis. Intensive Care Med. 2017 Feb;43(2):155-170. doi: 10.1007/s00134-016-4573-3. Epub 2016 Oct 12. PMID 27734109
- [Background] Salahuddin N, Sammani M, Hamdan A, Joseph M, Al-Nemary Y, Alquaiz R, Dahli R, Maghrabi K. Fluid overload is an independent risk factor for acute kidney injury in critically Ill patients: results of a cohort study. BMC Nephrol. 2017 Feb 1;18(1):45. doi: 10.1186/s12882-017-0460-6. PMID 28143505
- [Background] Bihari S, Prakash S, Potts S, Matheson E, Bersten AD. Addressing the inadvertent sodium and chloride burden in critically ill patients: a prospective before-and-after study in a tertiary mixed intensive care unit population. Crit Care Resusc. 2018 Dec;20(4):285-293. PMID 30482136
- [Background] Magee CA, Bastin MLT, Laine ME, Bissell BD, Howington GT, Moran PR, McCleary EJ, Owen GD, Kane LE, Higdon EA, Pierce CA, Morris PE, Flannery AH. Insidious Harm of Medication Diluents as a Contributor to Cumulative Volume and Hyperchloremia: A Prospective, Open-Label, Sequential Period Pilot Study. Crit Care Med. 2018 Aug;46(8):1217-1223. doi: 10.1097/CCM.0000000000003191. PMID 29727367
- [Background] Van Regenmortel N, Langer T, De Weerdt T, Roelant E, Malbrain M, Van den Wyngaert T, Jorens P. Effect of sodium administration on fluid balance and sodium balance in health and the perioperative setting. Extended summary with additional insights from the MIHMoSA and TOPMAST studies. J Crit Care. 2022 Feb;67:157-165. doi: 10.1016/j.jcrc.2021.10.022. Epub 2021 Nov 17. PMID 34798374
- [Background] Nagae M, Egi M, Furushima N, Okada M, Makino S, Mizobuchi S. The impact of intravenous isotonic and hypotonic maintenance fluid on the risk of delirium in adult postoperative patients: retrospective before-after observational study. J Anesth. 2019 Apr;33(2):287-294. doi: 10.1007/s00540-019-02626-4. Epub 2019 Feb 26. PMID 30806785
- [Background] Surveillance report 2017 - Intravenous fluid therapy in adults in hospital (2013) NICE guideline CG174 [Internet]. London: National Institute for Health and Care Excellence (NICE); 2017 Apr 24. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK552079/ PMID 31891467
- [Background] Haines RW, Zolfaghari P, Wan Y, Pearse RM, Puthucheary Z, Prowle JR. Elevated urea-to-creatinine ratio provides a biochemical signature of muscle catabolism and persistent critical illness after major trauma. Intensive Care Med. 2019 Dec;45(12):1718-1731. doi: 10.1007/s00134-019-05760-5. Epub 2019 Sep 17. PMID 31531715
- [Background] Kitada K, Daub S, Zhang Y, Klein JD, Nakano D, Pedchenko T, Lantier L, LaRocque LM, Marton A, Neubert P, Schroder A, Rakova N, Jantsch J, Dikalova AE, Dikalov SI, Harrison DG, Muller DN, Nishiyama A, Rauh M, Harris RC, Luft FC, Wassermann DH, Sands JM, Titze J. High salt intake reprioritizes osmolyte and energy metabolism for body fluid conservation. J Clin Invest. 2017 May 1;127(5):1944-1959. doi: 10.1172/JCI88532. Epub 2017 Apr 17. PMID 28414295
- [Background] Rakova N, Kitada K, Lerchl K, Dahlmann A, Birukov A, Daub S, Kopp C, Pedchenko T, Zhang Y, Beck L, Johannes B, Marton A, Muller DN, Rauh M, Luft FC, Titze J. Increased salt consumption induces body water conservation and decreases fluid intake. J Clin Invest. 2017 May 1;127(5):1932-1943. doi: 10.1172/JCI88530. Epub 2017 Apr 17. PMID 28414302

DOCUMENTS (4):
  • Study Protocol (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT07189091/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT07189091/SAP_001.pdf
  • Informed Consent Form: CRUSADERS main trial (2025-03-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT07189091/ICF_002.pdf
  • Informed Consent Form: SALADIN nested substudy (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT07189091/ICF_003.pdf